CLINICAL TRIAL: NCT04722783
Title: Effect of Early Start Denver Model and Autism-adapted Parent-Child Interaction Therapy on Autism Symptoms and Disruptive Behavior in Toddlers and Preschool Children with Autism Spectrum Disorder (TAFF Pilot Study)
Brief Title: Effect of ESDM and PCIT-A in Autism Spectrum Disorder
Acronym: TAFF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The final study period was 1 year longer than anticipated but only 24 instead of 28 participants could be included. In the context of resource limitations and a sufficient sample size to assess the study aims, we prematurely stopped the pilot trial.
Sponsor: Bruno Rhiner (Other)
Collaborators: West Virginia University (Other); University of Arkansas (Other)
Responsible Party: Sponsor-Investigator, Bruno Rhiner, Head of Child and Adolescent Psychiatry, Psychiatrische Dienste Thurgau
Organization: Psychiatrische Dienste Thurgau (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol_PDT_010_TAFF; 2020-02787 (EKOS 20/223) (Other: Ethics Committee of Eastern Switzerland (EKOS))
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Parent-Child Interaction Therapy; Early Start Denver Model; Autism Spectrum Disorder; Disruptive behavior; Autism Symptoms; Toddlers; Preschool children
MeSH Terms: conditions — Autism Spectrum Disorder; Problem Behavior | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a pilot, practical clinical trial with a single-blind, mixed randomized and non-randomized controlled factorial design within a monocentric setup
Who Masked: Outcomes Assessor
Masking Description: The DPICS rating - as part of the primary outcome - is the only measure that is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ESDM and PCIT-A (Experimental): Participants in this arm receive 2 years ESDM and after 4 months PCIT-A for 8 months (see Study Protocol, Figure 2).
  Interventions: Behavioral: Parent-Child-Interaction Therapy adapted for children with autism spectrum disorder (PCIT-A); Behavioral: Early Start Denver Model (ESDM) intervention
- ESDM and active control for PCIT-A (Experimental): Participants in this arm receive 2 years ESDM and after 4 months 1h-ESDM as active control instead of 1h-PCIT-A for 8 months
  Interventions: Behavioral: Early Start Denver Model (ESDM) intervention; Behavioral: 1-hour ESDM
- PCIT-A and active control for ESDM (Experimental): Participants receive after 4 month PCIT-A for 8 months and early special needs education as an active control for ESDM.
  Interventions: Behavioral: Parent-Child-Interaction Therapy adapted for children with autism spectrum disorder (PCIT-A); Behavioral: Early special needs education (ESNE)
- Active control for ESDM and PCIT-A (Active Comparator): Participants receive early special needs education as an active control for ESDM and PCIT-A.
  Interventions: Behavioral: Early special needs education (ESNE)

INTERVENTIONS:
Behavioral: Parent-Child-Interaction Therapy adapted for children with autism spectrum disorder (PCIT-A) — PCIT is a behavioral family therapy approach emphasizing the integration of traditional child play therapy techniques within a behavioral framework of parent-child therapy and was developed by Eyberg (1988). It is based on attachment theory, social learning theory, and parenting styles theory. Recently, the intervention was adapted to children with ASD by our team (McNeil, Quetsch, & Anderson, 2019). PCIT-A will last about 8 months, 1 day per week, 60min per day (see Study Protocol, Fig. 2).
  Other Names: Intervention I
  Arms: ESDM and PCIT-A; PCIT-A and active control for ESDM
Behavioral: Early Start Denver Model (ESDM) intervention — ESDM intervention provides intensive teaching by trained therapists and parents during natural play and relationship-focused daily routines. It is evidence-based and uses principles of developmental psychology and applied behavior analysis. It was designed for toddlers and preschoolers with autism spectrum disorder by Rogers and Dawson (2010). The first intensive part of ESDM intervention (20h per week) will last 40 weeks of intervention within a period of 12 months. It includes 2 days per week for 6h a day clinic therapy, and 5 days per week for 1h homework tasks, and 2 days per week for 1.5h an early special needs education at home. After the first 12 months, children receive the second lower intensity part of ESDM (7 hours per week). It includes 1 days every two weeks 1h day clinic therapy, and 5 days per week for 1h homework tasks, and 1 days per week for 1.5h an early special needs education at home (see Study Protocol, Fig. 2).
  Other Names: Intervention II
  Arms: ESDM and PCIT-A; ESDM and active control for PCIT-A
Behavioral: 1-hour ESDM — The active control group for PCIT-A stays in the ESDM day clinic therapy for the 12 hours per week while the PCIT-A group will receive 11 hours of ESDM day clinic therapy and 1 hour PCIT-A per week (see Study Protocol, Fig. 2).
  Other Names: Active control for Intervention I
  Arms: ESDM and active control for PCIT-A
Behavioral: Early special needs education (ESNE) — The wait-list control group will receive early special needs education. It consists of a 90-minute visit at participants' homes once a week by an employee educated in early special needs education. As soon as space in ESDM is available children will receive the ESDM intervention (stepped-wedge design, see Study Protocol, Fig. 2).
  Other Names: Active control for Intervention II
  Arms: Active control for ESDM and PCIT-A; PCIT-A and active control for ESDM

SUMMARY:
Children with ASD often show disruptive behaviors. However, interventions that were specifically designed to improve these symptoms have not been sufficiently investigated, especially in children with level 1 to level 3 ASD. PCIT has large effects on externalizing behavior problems in children with disruptive behavior disorders. Recently PCIT was adapted for children with autism spectrum disorder (PCIT-A). ESDM is an evidence-based treatment for ASD but has not been investigated in combination with PCIT-A.

As primary aims, the investigators assess a) the effect of PCIT-A on disruptive behavior and b) the effect of ESDM on autism symptoms in toddlers and preschool children with ASD level 1 to 3. As secondary aims, the investigators evaluate a) the maintenance of the effect of PCIT-A one year after the end of intervention and b) the effect of both interventions on secondary outcomes (developmental level, intelligence, adaptive behavior, and parenting stress), c) the combined intervention effect of PCIT-A and ESDM depending on intervention overlap periods.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a life-long neurodevelopmental disorder with recognizable symptoms often beginning between one and two years of age and an estimated prevalence of about 0.6%. Both social communication deficits, and restrictive and repetitive behavior depict the core symptoms of ASD.

ESDM is an evidence-based treatment for ASD. A recent meta-analysis comprising 12 studies show favorable effects of ESDM on cognition and language with a moderate effect size, in contrast to control groups. ESDM showed to become cost-efficient within a few years after treatment as a result of less use of other health care services in the years following the intervention.

Children with ASD often show disruptive behaviors such as angry outbursts, irritability, aggressive and oppositional behaviors. However, interventions that were specifically designed to improve these symptoms have not been sufficiently investigated, especially in children with level 1 to level 3 ASD. PCIT has large effects on externalizing behavior problems in children with disruptive behavior disorders. Recently, PCIT was adapted for children with autism spectrum disorder (PCIT-A).

As primary aims of the so-called TAFF (Tagesklinik für Autismus und Frühförderung [Day Clinic for Autism and Early Intervention]) pilot study, the investigators assess a) the effect of PCIT-A on disruptive behavior and b) the effect of ESDM on autism symptoms in toddlers and preschool children with ASD level 1 to 3. As secondary aims, the investigators evaluate a) the maintenance of the effect of PCIT-A one year after the end of intervention and b) the effect of both interventions on secondary outcomes (developmental level, intelligence, adaptive behavior, and parenting stress), c) the combined intervention effect of PCIT-A and ESDM depending on intervention overlap periods.

ELIGIBILITY:
Inclusion Criteria:

* ASD level 1 to 3
* Time commitment of at least one parent (including homework and traveling time)
* Willingness of one parent to be the study informant over the whole study period

Exclusion Criteria:

* Insufficient German language skills of both parents to participate in the intervention
* Severe hearing or visual impairment
* Attention deficit hyperactivity disorder
* Epilepsy
* Rett syndrome
* Other rare, severe neurological disorders that interfere with therapy

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Disruptive behavior change (for PCIT-A analysis) | Between 4-month and 12-month FU
  Change from 4-month to 12-month Follow-Up (FU) in a composite score of Dyadic Parent-Child Interaction Coding System percentage compliance score and Eyberg Child Behavior Inventory intensity score (objective and parent-reported disruptive behavior; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a worse outcome)
Autism symptoms change (for ESDM analysis) | Between baseline to 4 month FU
  Change from baseline to 4-month FU in Quantitative Checklist for Autism in Toddlers score (parent-reported, range: 0-100 points; higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Disruptive behavior long-term change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 24-month FU in a composite score of Dyadic Parent-Child Interaction Coding System percentage compliance score and Eyberg Child Behavior Inventory intensity score (objective and parent-reported disruptive behavior; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a worse outcome)
Autism symptoms change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 12-month FU and to 24-month FU in Quantitative Checklist for Autism in Toddlers score (parent-reported, range: 0-100 points; higher scores mean a worse outcome)
Developmental level change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 12-month and to 24-month FU in Entwicklungstest für Kinder von 6 Monaten bis 6 Jahren (engl.: Developmental Test for Children from 6 months to 6 years; behavioral and parent-reported measure, composite score of all 6 domains; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Non-verbal Intelligence change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 12-month and to 24-month FU in Snijders-Oomen Non-verbal intelligence test revised 2-8 - puzzle subtest; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Adaptive behavior change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 12-month and to 24-month FU in Vineland Adaptive Behavior Scale (composite score of the three domains communication, daily living skills, socialization; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Social-emotional competence change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 12-month and to 24-month FU in Devereux Early Childhood Assessment (18 to 36 months version; (composite score of the three domains attachement/relationships, initiative, self-regulation; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Parenting stress change (for PCIT-A analysis) | Between 4-month and 24-month FU
  Change from 4-month to 12-month FU and to 24-month FU in Eltern-Belastungs-Inventar (engl.: Parenting Stress Index; composite score of 12 subscales, z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a worse outcome)
Autism symptoms long-term change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 12-month FU in Quantitative Checklist for Autism in Toddlers score (parent-reported, range: 0-100 points; higher scores mean a worse outcome)
Disruptive behavior change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 4-month FU and from baseline to 12-month FU in a composite score of Dyadic Parent-Child Interaction Coding System percentage compliance score and Eyberg Child Behavior Inventory intensity score (objective and parent-reported disruptive behavior; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a worse outcome)
Developmental level change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 4-month FU and from baseline to 12-month FU in Entwicklungstest für Kinder von 6 Monaten bis 6 Jahren (engl.: Developmental Test for Children from 6 months to 6 years; behavioral and parent-reported measure, composite score of all 6 domains; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Non-verbal intelligence change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 4-month FU and from baseline to 12-month FU in Snijders-Oomen Non-verbal intelligence test revised 2-8 - puzzle subtest; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Adaptive behavior change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 4-month FU and from baseline to 12-month FU in Vineland Adaptive Behavior Scale (composite score of the three domains communication, daily living skills, socialization; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Social-emotional competence change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 4-month FU and from baseline to 12-month FU in Devereux Early Childhood Assessment (18 to 36 months version; (composite score of the three domains attachement/relationships, initiative, self-regulation; z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a better outcome)
Parenting stress change (for ESDM analysis) | Between baseline and 12-month FU
  Change from baseline to 4-month FU and from baseline to 12-month FU in Eltern-Belastungs-Inventar (engl.: Parenting Stress Index; composite score of 12 subscales, z-standardized values with mean of 0 and SD of 1; probable range between -3 and +3; higher scores mean a worse outcome)

OTHER OUTCOMES:
Disruptive behavior change within the PCIT-A subsample | Between 4-month and 24-month FU
  Change from 4-month to 24-month FU in disruptive behavior composite score (see primary outcome for a detailed description) depending on ESDM/PCIT-A intervention overlap
Autism symptoms change within the subsample that started with the ESDM intervention | Between baseline and 24-month FU
  Change from first to last session of the ESDM intervention in the Early Start Denver Model checklist (trainer-rating)
Age-standardized long-term effect in all outcomes within the ESDM/PCIT-A subsample | Between baseline and 24-month FU
  Age-standardized changes from baseline to 24-month FU in all outcomes with available age-norms within the subsample that started both interventions (PCIT-A and ESDM; age-standardized z-scores with mean of 0 and SD of 1; probable range between -3 and +3;higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Rhiner, Dr med, Principal Investigator — Psychiatric Services of Thurgovia
Locations (1):
- Psychiatric Services of Thurgovia, Münsterlingen, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided because of ethical considerations